CLINICAL TRIAL: NCT06310252
Title: A Prospective Multicenter Clinical Study to Evaluate the Safety and Effectiveness of Intrastromal Implantation of the Transform Corneal Allograft (TCA) for Providing Near Vision in Presbyopic Subjects - Long Term Follow-up
Brief Title: Safety and Efficacy of an Intrastromal Transform Corneal Allograft (TCA) for Presbyopia Correction - Long Term Follow-up
Status: Completed | Type: Observational
Sponsor: Allotex, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO_010-2023
Record Dates: First submitted 2024-02-29; First posted 2024-03-15 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Opthalmic assessments — The participants will undergo the following assessments:
  1. Pupil size measurement
  2. Manifest refraction (no autorefraction)
  3. Monocular in both eyes and binocular uncorrected visual acuity (photopic):
     * Distance (4 m)
     * Intermediate (80 cm)
     * Near (40 cm)
  4. Monocular best corrected visual acuity (photopic):
     * Distance (4 m)
     * Near (40 cm)
     * Distance-corrected near (40 cm)
  5. Monocular and binocular mesopic (with and without glare) and photopic (without glare) contrast sensitivity testing (subgroup)
  6. Slit lamp examination
  7. Tear breakup time
  8. Placido Corneal topography, keratometry and pachymetry
  9. Optical coherence tomography including epithelium mapping (subgroup)
  10. Applanation intraocular pressure
  11. Cycloplegic refraction
  12. Dilated fundus examination
  13. Wavefront aberrometry (subgroup)
  14. Adverse events

SUMMARY:
The objective of this clinical study is to evaluate the long term safety and effectiveness of intrastromal implantation of the Allotex TransForm corneal allograft (TCA) for providing near vision in presbyopic subjects.

A maximum of 101 eyes of qualified and consented subjects will undergo long term follow-up after instrastromal implantation of the TCA for presbyopia.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent, have signed the written informed consent form, and been given a copy.
* Subjects must be willing and able to return for one scheduled follow-up examinations.
* Subjects must have undergone implantation with the TCA under study protocol PRO-010 between April 24, 2019 and October 31, 2019.

Exclusion Criteria:

• There are no known exclusion criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A maximum of 101 eyes of qualified and consented subjects will undergo long term follow-up after instrastromal implantation of the TCA for presbyopia.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2024-02-13 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
An exploratory data collection project with no primary safety or effectiveness endpoints. | 4 years or more after TCA implantation
  An exploratory data collection project with no primary safety or effectiveness endpoints.

CONTACTS AND LOCATIONS:
Locations (7):
- Gemini - Oční klinika Zlín, Zlín, Czechia
- Wellington Eye Clinic, Dublin, Ireland
- Medipol University, Istanbul, Turkey (Türkiye)
- United Kingdom (4):
  - Centre For Sight, East Grinstead
  - Eye Clinic London, London
  - Centre For Sight, London
  - Centre For Sight, Oxshott